CLINICAL TRIAL: NCT03841487
Title: All-cause Mortality and the Risk of Stroke With Selective Aspiration Thrombectomy in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention - A Nationwide Retrospective Cohort Study
Brief Title: Selective Aspiration Thrombectomy in STEMI
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chang Tung, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: CMRPG3E1051
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST-elevation myocardial infarction; Thrombectomy; Mortality; Stroke; Physician volume
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Stroke | interventions — Thrombectomy; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspiration thrombectomy: In the aspiration thrombectomy group, aspiration thrombectomy was performed for patients with ST elevation myocardial infarction who underwent primary percutaneous coronary intervention (PCI).
  Interventions: Device: Aspiration thrombectomy
- PCI alone: In the PCI alone group, the STEMI patient received conventional primary PCI without aspiration thrombectomy during the procedure.

INTERVENTIONS:
Device: Aspiration thrombectomy — In the aspiration thrombectomy group, aspiration thrombectomy was performed for patients with ST elevation myocardial infarction who underwent primary percutaneous coronary intervention (PCI). In the PCI alone group, the STEMI patient received conventional primary PCI without aspiration thrombectomy during the procedure.
  Other Names: Percutaneous coronary intervention
  Groups: Aspiration thrombectomy

SUMMARY:
Patients who were diagnosed with ST-elevation myocardial infarction (STEMI) and received primary percutaneous coronary intervention (PPCI) from July 2009 to December 2011 were identified from the National Health Insurance Research Database of Taiwan. The investigators compared the 1-year outcomes of patients with STEMI who received aspiration thrombectomy during PPCI vs. those who received PPCI alone.

DETAILED DESCRIPTION:
Data source and study population Using the National Health Insurance Research Database of Taiwan, STEMI patients from July 2009 to December 2011 who received aspiration thrombectomy during PPCI were defined as the thrombectomy group, and the remaining patients were defined as the PCI alone group. ICD-9-CM codes were used to identify underlying comorbidities. Data regarding the prescription of in-hospital and outpatient medications and the utilization of medical devices were also extracted from the NHIRD using ICD-9-CM procedure codes and pharmacology and device codes.

Study outcomes The primary endpoints of this study were all-cause mortality and stroke during hospitalization and at 30 days and 1 year of follow-up. Ischemic and hemorrhagic subtypes of stroke were further identified according to ICD-9-CM codes. All patientswere followed for 1 year or until the outcomes were achieved, whichever came first.

Statistical analysis Propensity score weighting was used to reduce potential differences between the two study groups. The incidence rates of all-cause mortality and stroke were estimated as the total number of events during the follow-up period divided by the person-months at risk. For all-cause mortality, a Cox proportional hazard model was used to obtain hazard ratios (HRs). For stroke, Fine and Gray's competing-risk regression was used to obtain sub-hazard ratios (SHRs). The cumulative incidence of stroke versus follow-up time was plotted rather than the event-free rate, because cumulative incidence function can take the competing risk of death into account. For the thrombectomy group, 95% confidence intervals (CIs) of the HRs and SHRs were calculated using the PCI alone group as the referent group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST elevation myocardial infarction

Exclusion Criteria:

* Missing data on sex or discharge date
* Aged less than 18 years
* Previous stroke
* Patients receiving thrombolytic therapy
* Patients who did not undergo PPCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ST elevation myocardial infarction who received primary percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 9100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of all-cause mortality at 30 days | 30 days from the date of primary percutaneous coronary intervention
  The total number of death during the follow-up period divided by the person-months at risk
Incidence rate of stroke at 30 days | 30 days from the date of primary percutaneous coronary intervention
  The total number of stroke events during the follow-up period divided by the person-months at risk
Incidence rate of all-cause mortality at 1 year | 1 year from the date of primary percutaneous coronary intervention
  The total number of death during the follow-up period divided by the person-months at risk
Incidence rate of stroke at 1 year | 1 year from the date of primary percutaneous coronary intervention
  The total number of stroke events during the follow-up period divided by the person-months at risk

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chang Tung, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data is encrypted and is not allowed to share based on the regulations of the National Health Insurance Research Database of Taiwan.